CLINICAL TRIAL: NCT07351292
Title: Comparative Study of Therapeutic Ultrasound and Whole-body Vibration as Adjuncts to Passive Stretching on Knee Joint Range of Motion and Functional Ability in Children With Hemiplegic Cerebral Palsy.
Brief Title: Ultrasound or Whole Body Vibration on Knee Motion and Function in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa S Ali, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006029
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP)
Keywords: Ultrasound; whole-body vibration; knee range of motion; functional ability; children; hemiplegia; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Investigator
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound group (Experimental): received therapeutic ultrasound prior to stretching
  Interventions: Device: ultrasound
- whole body vibration group (Experimental): performed exercises on a vibrating platform before stretching
  Interventions: Device: whole body vibration

INTERVENTIONS:
Device: ultrasound — Received continuous ultrasound (1 MHz, 1.0 W/cm², 5 min per hamstring) using a Chattanooga Intelect Mobile 2 unit with a medium-sized transducer head and coupling gel
  Arms: ultrasound group
Device: whole body vibration — Performed exercises on a Power Plate Pro 5 vibration platform. Parameters were set to a frequency of 20 Hz and a fixed amplitude of 2 mm (peak-to-peak displacement). The child maintained a semi-squat posture (approximately 30 knee flexion) for two 5-minute bouts separated by a 1-minute rest.
  Arms: whole body vibration group

SUMMARY:
This study compared the efficacy of therapeutic ultrasound (US) and whole-body vibration (WBV) as adjuncts to a standardized passive stretching regimen on improving knee joint range of motion (ROM) and functional capacity in children with hemiplegic cerebral palsy (HCP).

DETAILED DESCRIPTION:
Sixty children with HCP, aged 4-6 years, were randomly assigned to one of two groups. Both groups received passive stretching of the hamstrings and plantar flexors three times per week for twelve weeks. The control group (US group) received therapeutic ultrasound prior to stretching, while the research group (WBV group) performed exercises on a vibrating platform before stretching. Active knee extension ROM was measured with a digital goniometer, and functional ability was assessed using the Gross Motor Function Measure-88 (GMFM-88) at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* age from 4-6 years
* knee flexion deformity due to hamstring tightness
* Gross Motor Function Classification System (GMFCS) levels I or II
* spasticity grade of 1 or 2 on the modified Ashworth Scale

Exclusion Criteria:

* other causes of knee flexion deformity
* previous orthopedic knee surgery
* significant visual, auditory, or perceptual deficits
* uncontrolled seizures; or acute illness

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Range of Motion (ROM) | 12 weeks
  Measured using an Absolute + Axis™ Digital Goniometer. With the child supine and pelvis stabilized, the goniometer axis was aligned with the lateral femoral condyle. The stationary arm was aligned with the greater trochanter, and the moving arm with the lateral malleolus. The child was instructed to actively extend the knee as far as possible, and the angle was recorded. Three measurements were taken, and the average was used for analysis
2. Gross Motor Function | 12 weeks
  Assessed using the Gross Motor Function Measure-88 (GMFM-88), a validated observational tool for children with CP. A blinded assessor, not involved in the intervention, scored the children's performance. The Gross Motor Functional Measurement-88 used to measure function. The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline. However, most of the items have specific descriptors for each score. It is imperative that the guidelines
  contained in the manual be used for scoring each item.
  SCORING KEY 0 = does not initiate
  1. = initiates
  2. = partially completes
  3. = completes

CONTACTS AND LOCATIONS:
Overall Officials: mostafa S ali, PhD, Principal Investigator — associate professor for pediatrics
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided